CLINICAL TRIAL: NCT04121377
Title: Feasibility of an Early Progressive Strength Exercise Programme for Acute Achilles Tendon Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Christensen, PT, PHD student, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20180072
Record Dates: First submitted 2019-09-29; First posted 2019-10-09 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Achilles Tendon Rupture
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance exercise program (Experimental): Early resistance exercise sessions and home program
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — Weekly sessions introducing resistance exercises and monitoring the patients acceptability. The exercises are isometric contractions, seated heel-rise and elastic band. The patient register the amount of exercise in a home exercise journal. To protect the tendon while doing range of motion of the foot, dorsiflexion is restricted beyond neutral (0 degrees of dorsiflexion). The load on the strength exercises will progress from isometric contraction without external load to strengthening exercises with 10-20 RM (RM: Repetition Maximum). Each strength exercise can progress with added weight or stronger elastic band. The Borg scale is used to guide the patient to progress or regress the load in each exercise. The recommended level being "easy" to "hard" (2-5/10). It is emphasised that the exercises must not cause sudden or severe pain in the tendon, but muscle soreness is to be expected.

SUMMARY:
The aim of this study is to investigate the feasibility of an early progressive exercise program for patients with Achilles tendon rupture treated non-surgically. The outcomes will concern the patient's acceptability of the intervention, adherence to the intervention and safety of the healing tendon.

DETAILED DESCRIPTION:
Regardless of choice of either surgical or non-surgical treatment, long-term muscular deficits and a decreased function after Achilles tendon rupture is found up to 10 years later. The majority of the patients are of working age and a deficit in physical performance will have impact on returning to work and sports.

There has been promising results in treatments using early functional rehabilitation during the first eight weeks of treatment after both surgical and non-surgical treatment, but few studies has examined the effect of the exercises on its own. In general, descriptions of the exercise programs are lacking important information such as type, time of application, frequency, intensity and progression of the exercises.

The primary aim is to test the feasibility of an early progressive exercise program for patients with Achilles tendon rupture treated non-surgically. Feasibility in this study will be defined as successful patient acceptability and compliance of the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Acute Achilles tendon rupture treated non-surgically
* Diagnosed and treatment initiated within 3 days of injury
* Age 18-65, able and willing to participate in the intervention
* Able to speak and understand Danish

Exclusion Criteria:

* Insertional Achilles tendon rupture on calcaneus or rupture in the musculo-tendinous junction of the triceps surae
* Previous Achilles tendon rupture or other conditions in either leg causing lower leg disability (pain, deficits in strength or range of movement)
* Treated with Fluoroquinolones or Corticosteroids within the last 6 months
* Diabetes
* Severe medical illness: ASA score higher than or equal to 3. (ASA: American Society of Anesthesiologists physical status classification system)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | At 10 week follow-up
  The participants will rate their acceptability (willingness) to perform the exercises on a 7-point Likert scale ranging from "very unacceptable" to "very acceptable". This is not a measure of whether the patient's symptoms have improved to normal physical function or any other satisfactory level at the specific time, but if it matches, their expectations of the content of an exercise program in this early phase and how they tolerate performing the exercises. The intervention program is categorised as "Unacceptable" if rated as the three lower scores ("very unacceptable" to "slightly unacceptable") and categorised as "Acceptable" if rated as the four higher scores ("neither acceptable or unacceptable" to "very acceptable"). The exercise program is considered feasible if acceptability of the exercise program is 80%. Defined as: ≥13/16 patients will rate the acceptability of the intervention as "acceptable".
Compliance | At 10 week follow-up
  The participants will register the number of training sessions and exercises they perform each day in a training journal. The compliance is measured as the mean number of exercise sessions they perform. The timeframe will be from the day they start the exercises to the end of week 9. The exercise program is considered feasible if the adherence to the exercise program is 50%. Defined as: ≥13/16 patients will perform ≥ 50% of the exercise sessions possible from start to end of week 9.

SECONDARY OUTCOMES:
Fear of re-rupture | At 2 and 10 weeks and at 3 months
  The Tampa scale of Kinesiophobia (TSK) is a questionaire consisting of 17 items concerning pain and kinesiophobia and has 4 answers from "Strongly disagree" to "Strongly agree". During the exercise intervention period and at 3 months follow,up the patients will fill out the score and subsequently they are asked to rate the appropriateness of the score on a 7 point Likert scale ranging from "strongly disagree" to "strongly agree".
Achilles tendon total rupture score (ATRS) | Baseline for a pre-rupture level and at 3 months
  Validated patient reported outcome measure. It contains 10 questions about physical performance in an 11-point Likert scale from zero to ten.
Physical Activity | Baseline for a pre-rupture level and at 3 months
  International Physical Activity Questionnaire (IPAQ) short form Danish version. It consists of 7 items concerning physical activity as time spent performing vigorous and moderate activities, the time spent walking and sitting during the past week. The IPAQ gives an estimate of the total weekly physical activity measured in MET-minutes per week and total minutes spent sitting.(MET: The Metabolic Equivalent of Task)
Achilles tendon resting angle (ATRA) | At 10 weeks and at 3 months
  Indirect measure of the Achilles tendon length. It is measured in degrees between the axis of the fibula (from malleol to proximal head) and the line from the tip of the fibula to the head of the Fifth metatarsal bone.
Achilles tendon length | At 10 weeks and 3 months
  Ultrasound measure of achilles tendon length.,
Achilles tendon cross-sectional area | At 10 weeks and 3 months
  Ultrasound measure of cross-sectional area of the Achilles tendon at the rupture site
Delay in start of exercise | At 10 weeks
  Delay in starting the exercise program is measured in days drom start to end of week 9
Adverse events | At 10 weeks and 3 months
  The number of serious and minor adverse events is registered using open questions and a pre-defined list.
Muscle endurance | At 3 months
  Muscle endurance is measured in seated heel-rise with MuscleLab Measurement system (Ergotest Technology, Oslo, Norway)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Christensen, MHSc, Principal Investigator — Physiotherapy and Occupational Therapy, Aalborg University Hospital
Locations (1):
- Physiotherapy and Occupational Therapy, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request

REFERENCES:
- [Derived] Christensen M, Silbernagel KG, Zellers JA, Kjaer IL, Rathleff MS. Feasibility of an early progressive resistance exercise program for acute Achilles tendon rupture. Pilot Feasibility Stud. 2024 Apr 22;10(1):66. doi: 10.1186/s40814-024-01494-4. PMID 38650039

DOCUMENTS (1):
  • Study Protocol (2019-09-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT04121377/Prot_000.pdf